CLINICAL TRIAL: NCT00701454
Title: Survey of Thai-Muslim Health Status
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Nipa Rojroongwasinkul / Assistant Professor, Institute of Nutrition, Mahidol University
Other Study IDs: INMU-2006-01
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes; Hypertension; Hyperlipidemia
Keywords: Thai-muslim; Thai-HALAL; Diabetes; Hypertension; Hyperlipidemia; Metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy participants (physically and mentally).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study was to determine the prevalence and risk factors of diabetes, hypertension, hyperlipidemia among Thai muslim population aged 35-75 years.

DETAILED DESCRIPTION:
This was a cross-sectional study conducted in Bangkok and surrounding provinces. Approximately 1500 participants were enrolled. Study staff interviewed participants on basic demographic data, health status, physical activities, food frequency and 24-hour recall. Anthropometry (body weight, height, hip and waist circumference) and physical assessment (blood pressure)were measured. Ten milliliters of venous blood was drawn by venipuncture after a 12 h overnight fast for determination of fasting plasma glucose (FPG) and blood lipid concentrations (total cholesterol, triglyceride, and HDL-cholesterol). FPG was measured by the enzymatic colorimetric method with glucose oxidase.21 Total cholesterol was determined by the cholesterol oxidase method and serum triglycerides concentration was determined by standardized enzymatic procedures using glycerol phosphate oxidase assay.22, 23 HDL- cholesterol was measured by enzymatic assays.24 LDL cholesterol was calculated according to the method of Friedwald et al.25 All samples were analyzed when internal quality control met the acceptable criteria. Intra-and inter-assay CVs were 2.01% and 3.01% for FPG, 1.87% and 4.24% for total cholesterol, 0.93% and 11.6% for triacylglycerols, and 0.99% and 1.49% for HDL cholesterol, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 35 y and older muslim
* free from severe communicable diseases and mental disorders

Exclusion Criteria:

* not able to complete the interviews or obtain blood samples for analysis

Ages: 35 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thai muslim residents in 4 muslim communities in and around Bangkok.
Sampling Method: Non-Probability Sample
Enrollment: 1488 (Actual)
Dates: Start 2005-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
prevalence of diabetes, hypertension and hyperlipidemia | after a 12 h overnight fast

CONTACTS AND LOCATIONS:
Overall Officials: Emorn Wasantwisut, Ph.D., Study Director — Mahidol University
Locations (1):
- Institute of Nutrition, Mahidol University, Phuttamonthon, Changwat Nakhon Pathom, Thailand